CLINICAL TRIAL: NCT05413096
Title: Combination of Diclofenac Potassium and Propolis in the Therapy of Oral Aphthosis
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Mohamed Ismail Assadawy, principle investigator, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: oral Aphthosis 650/3607
Record Dates: First submitted 2022-06-07; First posted 2022-06-09 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Oral Mucositis; ORAS; Oral Infection; Oral Ulcer
Keywords: diclofenac; oral disease; oral Aphthosis; propolis
MeSH Terms: conditions — Stomatitis; Oral Ulcer; Mouth Diseases | interventions — Propolis

STUDY DESIGN:
Intervention Model Description: A randomized clinical, double-blind, placebo-controlled study
Who Masked: Participant, Care Provider, Investigator
Masking Description: caregiver and participants and investigator are masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- placebo tube (Placebo Comparator): neutral material without any biological effects
  Interventions: Other: placebo
- Combination of diclofenac potassium and propolis (Active Comparator): active agents combination of diclofenac potassium 3% (10 mg/g, 60 g, EMS) and Propolis 5% gel
  Interventions: Combination Product: Combination of diclofenac potassium and propolis

INTERVENTIONS:
Combination Product: Combination of diclofenac potassium and propolis — Patients will be divided into two groups: the first one will be treated with a combination of diclofenac 3% (10 mg/g, 60 g, EMS) and Propolis 5% gel and the second one is placebo group. Participants will be allocated randomly. The patients will be asked to apply gel 2 times per day. The patients will be instructed, not to eat or drink for 1 h after application of the gel
  Arms: Combination of diclofenac potassium and propolis
Other: placebo — placebo
  Arms: placebo tube

SUMMARY:
The combination of diclofenac and propolis could enhance the healing of recurrent aphthous ulcers, instantly relieve symptoms, improve the quality of life, and present a de novo and cost-effective regime help in oral ulcer treatment. This study aimed to evaluate the influence of diclofenac and propolis combination as a gel in the treatment of recurrent oral ulceration

ELIGIBILITY:
Inclusion Criteria:

* patients have an oral mucosal ulcer

Exclusion Criteria:

* patients allergic to any component of the diclofenac formulation and other NSAIDs

Ages: 5 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
chronic oral mucosal disease questionnaire | 10 days
  patient response

SECONDARY OUTCOMES:
ulcer characters | 10 days
  size

CONTACTS AND LOCATIONS:
Locations (1):
- Al Azhar university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
individual participant data can be shared through the organization
Supporting Information: CSR
Time Frame: 6 months
Access Criteria: main investigator